CLINICAL TRIAL: NCT04105673
Title: Prognostic Factors for Sequelae in Children With a History of Shaken Baby Syndrome in the Central Region
Brief Title: Predictors of Sequelae Appearance in Shaken Baby Syndrome
Acronym: FPASSBS
Status: Withdrawn | Type: Observational
Why Stopped: CPP requalification
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18/FPASSBS; 2018-A03098-47 (Other: IdRCB)
Record Dates: First submitted 2019-01-11; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Shaken Baby Syndrome
Keywords: Shaken Baby Syndrome; long-term outcome; severity criteria in the admission to hospital for a Shaken Baby Syndrome; sequelae; brain injury; abusive head trauma
MeSH Terms: conditions — Shaken Baby Syndrome; Brain Injuries | interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shaken Baby Syndrome: Realization of a clinical examination and survey on children with a past history of a Shaken Baby Syndrome
  Interventions: Other: Clinical examination and survey

INTERVENTIONS:
Other: Clinical examination and survey — Children will be seen during an one consultation. A clinical examination and survey are realized.

SUMMARY:
This is an observational, prognostic and prospective study. It is about the Prognostic Factors for sequelae in children with a history of Shaken Baby Syndrome (SBS) in the Central region in France. The study hypothesis is the prognosis of the sequelae children develop according to the severity criteria presents in admission to the hospital for the Shaken Baby Syndrome. The severity criteria are clinical high intracranial pressure, presence of a coma, vitreous hemorrhage, an age under 6 months, other cerebral lesion than subdural hematoma (parenchymal lesion, ischemia or cerebral oedema). Children affected by the nonaccidental head injury are today between five and eight years old.

DETAILED DESCRIPTION:
Abusive head trauma is a severe inflicted traumatic brain injury, occuring under the age of 1 year, defined by an acute brain injury (mostly subdural or subarachnoidal haemorrhage), where no history or no compatible history with the clinical presentation is given.

This is secondary to violent shaking, with or without impact, of an infant by an adult, sufficient to cause brain injury. The mortality rate is estimated at 20-25% and growth of child is extremely poor. High rates of impairment are reported : motor deficit (spastic hemiplegia or quadriplegia), epilepsy often intractable, microcephaly with corticosubcortical atrophy, visual impairment even the blindness, language disorders, cognitive (intellectual deficit), behavioral (agitation, aggression, attention deficit, inhibition deficit) and sleep disorders. Several studies on the subject highlighted that an initial severe presentation is associated with worse growth.

These is very limited research on the outcome of inflicted traumatic brain injury and the results are heterogeneous. The study hypothesis is the prognosis of the sequelae children develop according to the severity criteria presented in admission to the hospital for the Shaken Baby Syndrome.

This is an epidemiological, observational, prognostic and prospective study. The severity criteria are clinical high intracranial pressure, presence of a coma, vitreous haemorrhage, an age under 6 months, other injuries than subdural hematoma (parenchymal injuries, ischemia or cerebral oedema).

The severity criteria were chosen by studying others studies on the subject. Children concerned had been admitted to hospital for Shaken Baby Syndrome between 2010 and 2014 in France, in the Central Region. Thus today, they are between five and eight years old. We know that sequelae occur after latency, in particular when children learn to read and write.

Primary purpose is to evaluate prognostic factors to develop sequelae after an inflicted traumatic brain injury as the shaken baby syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Children must be between five and eight years old
* Hospitalization before one year old for a Shaken Baby Syndrome in the Center Region in France

Exclusion Criteria:

* Opposition of the legal representative to use the data

Ages: 5 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: Children concerned had been admitted to hospital for Shaken Baby Syndrome before one year old in France, in the Central region
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
the sequelae motor developed by children with a past history of a Shaken Baby Syndrome. | At the inclusion (Day 1)
  The motor function is assessed by clinical neurological examination.
the cognitive sequelae developed by children with a past history of a Shaken Baby Syndrome | At the inclusion (Day 1)
  The cognitive function is assessed by the Wechler Scale (WPPSI IV). This scale assesses the verbal understanding, spatial visual understanding, fluid reasoning, work memory and treatment speed.
the behavioral sequelae developed by children with a past history of a Shaken Baby Syndrome. | At the inclusion (Day 1)
  Adaptive behavior is measured using the Vineland Adaptive Behavior Scales. This scale assesses 4 fields : communication, autonomy, socialization and motor function

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Saint Martin, MD-PhD, Study Director — University Hospital, Tours